CLINICAL TRIAL: NCT07171047
Title: Effects of Sodium Bicarbonate Supplementation on Endurance Performance and Physiological Responses During Simulated Cycling Competition
Brief Title: Effects of Sodium Bicarbonate on Endurance Performance
Acronym: SBEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salzburg (Other)
Collaborators: Red Bull Athlete Performance Center (Unknown)
Responsible Party: Principal Investigator, Nils Haller, PhD, Senior Researcher, University of Salzburg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BICARB_Haller
Record Dates: First submitted 2025-07-25; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Athlete; Well-trained Athletes; Performance
Keywords: Bicarbonate; Endurance training; Cycling; Time trial

STUDY DESIGN:
Intervention Model Description: Double blinded two-intervention crossover study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo then Verum (Other): Placebo then Verum 3 hour low-intensity ride followed by a 16 km time trial for both conditions. Supplementation of Placebo or Verum before the exercise start.
  Interventions: Dietary Supplement: Placebo then Verum
- Verum then Placebo (Other): Verum then Placebo 3 hour low-intensity ride followed by a 16 km time trial for both conditions. Supplementation of Placebo or Verum before the exercise start.
  Interventions: Dietary Supplement: Verum then Placebo

INTERVENTIONS:
Dietary Supplement: Placebo then Verum — Intake of 0.3 g/kg bodyweight of maltodextrin with hydrogel as placebo and 0.3 g/kg bodyweight of sodium bicarbonate with hydrogel as Verum
  Arms: Placebo then Verum
Dietary Supplement: Verum then Placebo — Intake of 0.3 g/kg bodyweight of maltodextrin with hydrogel as placebo and 0.3 g/kg bodyweight of sodium bicarbonate with hydrogel as Verum
  Arms: Verum then Placebo

SUMMARY:
This study is investigating whether taking sodium bicarbonate, a common supplement used by endurance athletes, can improve cycling performance during prolonged exercise and in a time trial. Sodium bicarbonate may help reduce muscle acidity, which could delay fatigue and improve performance. The goal of this study is to determine if this supplement can help athletes perform better during long, intense efforts like those seen in real competitions.

Participants in this study are well-trained cyclists who will complete two exercise trials in a laboratory setting. Each trial involves three hours of moderate cycling followed by a 20-30-minute time trial at maximum effort. Before each trial, participants will take either sodium bicarbonate or a placebo.

The study will measure performance outcomes, such as time trial results, as well as physiological responses, including heart rate, oxygen use, and muscle fatigue. Researchers hope to better understand how sodium bicarbonate can help endurance athletes and provide guidelines for its use in competitive sports.

ELIGIBILITY:
Inclusion Criteria:

* age 16-50 years
* well-trained cyclists
* Proof of physical fitness (e.g. sports medical examination required) for measurements with higher intensities (e.g. endurance tests, competition simulation)
* >10h endurance training per week

Exclusion Criteria:

* Systemic disease or other known pathology in the organs: heart, lungs, kidney, stomach, spleen, liver, gall bladder, and intestines.
* Evidence of pulmonary disease: forced expiratory volume in one second/forced expiratory volume < 70% with/without symptoms (cough, sputum) or other evidence of pulmonologic disease.

Diabetes II.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Endurance performance | 20-30 minutes, immediately after completion of the time trial for each condition (Placebo and Verum), assessed on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in time trial performance (average power in watts) between placebo and verum condition

SECONDARY OUTCOMES:
Difference in questionnaire score - gastrointestinal symptoms | 6.5 hours (rest, breakfast, every 30min during 3-hour low-intensity, after TT) for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in questionnaire score gastrointestinal symptoms between placebo and verum condition (0-10, higher score indicates more severe symptoms).
Difference in questionnaire score - Energy & Confidence | 3 hours (every 30min during 3-hour low-intensity) for each condition (Placebo and Verum), assessed on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in questionnaire score energy and confidence in time trial performance between placebo and verum condition (0-10, higher score indicates more Energy or Confidence in time trial performance).
Difference in questionnaire score - rate of perceived exertion | 3.5 hours (every 30min during 3-hour low-intensity, after TT) for each condition (Placebo and Verum), assessed on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in questionnaire score overall and legs only perceived exertion between placebo and verum condition (0-10, higher score indicates a higher degree of perceived exertion).
Difference in blood count | 6.5 hours (rest, every 30min during 3-hour low-intensity, after TT) for each condition (Placebo and Verum), assessed on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in capillary blood count between placebo and verum condition
Difference in pH & HCO3 kinetics | 6.5 hours (rest, breakfast, every 30min during 3-hour low-intensity, after TT) for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in pH & HCO3 kinetics between placebo, verum and resting verum condition
Difference in heart rate | 3.5 hours, assessed continuously (every second) during 3 hour low-intensity and TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in heart rate (bpm) between placebo and verum condition
Difference in oxygen uptake | 3 hours, assessed for 5 min every 30 min during 3 hour low-intensity for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in oxygen uptake (ml/kg/min) between placebo and verum condition
Difference in blood lactate concentration | 3.5 hours, assessed every 30 min during 3 hour low-intensity and after TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in blood lactate concentration (mmol/L) between placebo and verum condition.
Difference in substrate utilization | 3 hours, assessed for 5 min every 30 min during 3 hour low-intensity for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in substrate utilization between placebo and verum condition.
Difference in ventilation | 3 hours, assessed for 5 min every 30 min during 3 hour low-intensity for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in ventilation (L/min) between placebo and verum condition
Difference in core body temperature | 3.5 hours, assessed continuously during 3 hour low-intensity and TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in core body temperature (°) between placebo and verum condition.
Difference in muscle oxygenation | 3.5 hours, assessed continuously during 3 hour low-intensity and TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in muscle oxygenation (SmO2) of the vastus lateralis between placebo and verum condition.
Difference in glucose level | 24 hours, assessed continuously for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in glucose level (mg/dl) between placebo and verum condition.
Difference in sodium content | 3.5 hours, assessed during 3 hour low-intensity and TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in sodium content (mg/hr) between placebo and verum condition
Difference in sweat rate | 3.5 hours, assessed during 3 hour low-intensity and TT for each condition (Placebo and Verum), on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in sweat rate (L/hr) between placebo and verum condition.
Difference in next morning weight | 24 hours, assessed in the morning for each condition (Placebo and Verum) and the following day, on test day 1 and test day 2 respectively, with a washout period of 3-7 days between appointments (test days).
  Difference in weight (kg) measured in the morning of the test day and the following day (before breakfast after urination and defecation)

CONTACTS AND LOCATIONS:
Locations (1):
- Red Bull Athlete Performance Center, Thalgau, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided